CLINICAL TRIAL: NCT03752749
Title: Impact of Intermittent Hypoxia and Prednisolone on Motor Performance in Persons With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Zev Rymer, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00103487
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone + Acute Intermittent Hypoxia (Experimental)
  Interventions: Other: Prednisolone + Acute Intermittent Hypoxia
- Placebo + Acute Intermittent Hypoxia (Placebo Comparator)
  Interventions: Other: Placebo + Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Prednisolone + Acute Intermittent Hypoxia — Administration of oral prednisolone followed by 15, 60-second bouts of mild hypoxia
  Arms: Prednisolone + Acute Intermittent Hypoxia
Other: Placebo + Acute Intermittent Hypoxia — Administration of oral matching placebo followed by 15, 60-second bouts of mild hypoxia
  Arms: Placebo + Acute Intermittent Hypoxia

SUMMARY:
The objective of this study is to examine the effects of mild acute intermittent hypoxia (AIH) in combination with an anti-inflammatory drug (i.e. prednisolone) on motor performance in persons with spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord lesion at the level of C4 or below.
* Incomplete spinal cord injury ASIA (American Spinal Injury Association) Impairment Scale classification C or D. ASIA C or D classification requires that individuals have detectable motor function below the level of spinal injury and have preserved sensation of the sacral segments S4-S5 (anal sphincter).
* Age between 18 and 65 years.
* Medically stable with medical clearance to participate.
* SCI due to non-progressive etiology.
* More than 6 months since initial SCI. We plan to choose subjects greater that six months post-injury, to ensure minimal confounding effects of spontaneous neurological recovery during the experiments. This will mean that changes in motor performance are due to the interventions associated with the research study.
* Subjects must have active and passive ROM at the ankle from 10 degrees dorsiflexion to 30 degrees plantar flexion, 0 to 120 degrees of knee flexion, 90 degrees of hip flexion, and 10 degrees of hip extension in order to be positioned correctly for motor performance testing.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Presence of severe medical illness, including cardiac disease, uncontrolled high blood pressure, restrictive or obstructive pulmonary disease, significant osteoporosis or history of fracture following SCI, or history of lower limb peripheral nerve injury.
* Individuals with uncontrolled diabetes mellitus, unhealed decubitus ulcers, active heterotopic ossification, rheumatologic disease or inflammatory arthritis, presence of a deep venous thrombosis, cancer, or active infection will be excluded, as these conditions can cause systemic inflammation independent of spinal cord injury.
* Patients may not be receiving any other investigational agents.
* Individuals with tracheostomy, asthma, or recent or current pulmonary infection will be excluded.
* Women who are pregnant or nursing will be excluded, as the potential effects of intermittent hypoxia on pregnant women and fetus are unknown.
* Subjects will also be excluded if they are currently taking NSAIDs, steroids, or disease-modifying anti-rheumatic drugs (DMARDs). Participation is allowed if the subject and his/her physician agree to suspend all NSAIDs for a minimum of a 14-day washout period prior to study evaluation and for the duration of the study. Individuals taking oral steroids, DMARDs will be excluded from the study due to the potential risks of abruptly discontinuing these agents.
* Individuals will be excluded if they have a history of severe adverse reaction or allergic response to prednisolone in the past, history of stomach or intestinal ulcers, bleeding problems, chronic kidney disease, drink more than 3 alcoholic beverages per day, or are currently taking blood thinners. Excluding these individuals will limit the potential for having an adverse reaction to the anti-inflammatory administered in the study.
* Individuals receiving intrathecal baclofen will be excluded. Individuals prescribed medications other than intrathecal baclofen for alleviation of spastic motor behaviors will be excluded unless both the subject and his/her physician agree to cease all such medications for a 14-day minimum washout period prior to participation and for the duration of the study.
* Individuals will be excluded if they are taking antifungal ointments, estradiols or estrogens, rifampin, phenytoin, barbiturates or bupropion as these drugs can potential interact with prednisolone. See "concomitant medications" section below.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Isometric Ankle Plantar Flexion strength | 60 minutes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandhu MS, Gray E, Kocherginsky M, Jayaraman A, Mitchell GS, Rymer WZ. Prednisolone Pretreatment Enhances Intermittent Hypoxia-Induced Plasticity in Persons With Chronic Incomplete Spinal Cord Injury. Neurorehabil Neural Repair. 2019 Nov;33(11):911-921. doi: 10.1177/1545968319872992. Epub 2019 Sep 15. PMID 31524075